CLINICAL TRIAL: NCT02633527
Title: Evaluation of the Efficacy and Safety of SPN-812 (Viloxazine Extended-release Capsule) in Children With ADHD - A Double-Blind, Placebo-Controlled, Dose-Ranging Study
Brief Title: Efficacy and Safety of SPN-812 (Viloxazine Extended-release Capsule) in Children With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812P202
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2020-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Placebo (Placebo Comparator): Placebo, qd, oral capsule
  Interventions: Drug: Placebo
- 100mg SPN-812 (Experimental): 100mg SPN-812, qd, oral capsule
  Interventions: Drug: 100mg SPN-812
- 200mg SPN-812 (Experimental): 200mg SPN-812, qd, oral capsule
  Interventions: Drug: 200mg SPN-812
- 300mg SPN-812 (Experimental): 300mg SPN-812, qd, oral capsule
  Interventions: Drug: 300mg SPN-812
- 400mg SPN-812 (Experimental): 400mg SPN-812, qd, oral capsule
  Interventions: Drug: 400mg SPN-812

INTERVENTIONS:
Drug: Placebo — Placebo was administered once daily
  Other Names: PBO
  Arms: Placebo
Drug: 100mg SPN-812 — 100mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812, Low Dose
  Arms: 100mg SPN-812
Drug: 200mg SPN-812 — 200mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812, Low-Medium Dose
  Arms: 200mg SPN-812
Drug: 300mg SPN-812 — 300mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812, Medium-High Dose
  Arms: 300mg SPN-812
Drug: 400mg SPN-812 — 400mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812, High Dose
  Arms: 400mg SPN-812

SUMMARY:
This was a randomized, double-blind, placebo-controlled, multicenter, 5-arm, parallel-group, dose-ranging study to assess the efficacy and safety of SPN-812 (Viloxazine Extended-release Capsule) in children 6-12 years of age with ADHD.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multicenter, 5-arm, parallel-group, dose-ranging study to assess the efficacy, safety, and tolerability of SPN-812 (Viloxazine Extended-release Capsule) as monotherapy in the treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in children (6-12 years of age). Subjects are randomized in a 1:2:2:2:2 ratio to receive placebo or one of four active treatments (100 mg, 200 mg, 300 mg, or 400 mg SPN-812). The primary objective is to assess the efficacy of SPN-812 in reducing ADHD symptoms as measured by the Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, 6-12 years of age, inclusive, with a diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM IV), confirmed with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
2. ADHD-RS-IV-Parent Version: Investigator Administered and Scored score of at least 26.
3. CGI-S score of at least 4
4. Weight of at least 20 kg.
5. Free of medication for the treatment of ADHD or any psychosis for at least one week prior to enrollment.

Exclusion Criteria:

1. Current or lifetime diagnosis of major depressive disorder, bipolar disorder, personality disorder, Tourette's disorder, or psychosis not otherwise specified.
2. Currently meeting DSM-IV criteria for pervasive developmental disorder, obsessive compulsive disorder, post-traumatic stress disorder, or any other anxiety disorder as primary diagnosis.
3. Significant systemic disease.
4. Evidence of suicidality within the six months before Screening or at Screening.
5. BMI greater than 95th percentile for the appropriate age and gender.
6. Pregnancy or refusal to practice abstinence during the study for female subjects of childbearing potential (FOCP).
7. Substance or alcohol use during the last three months.
8. Positive urine screen for cotinine, alcohol, or drugs of abuse at Screening.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T. Hull, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (1):
- Florida Clinical Research Center, LLC, Maitland, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Treatment A: Placebo was administered once daily
- 100mg SPN-812: Treatment B: 100mg SPN-812 was administered once daily and compared to placebo
- 200mg SPN-812: Treatment C: 200mg SPN-812 was administered once daily and compared to placebo
- 300mg SPN-812: Treatment D: 300mg SPN-812 was administered once daily and compared to placebo
- 400mg SPN-812: Treatment E: 400mg SPN-812 was administered once daily and compared to placebo
Period: Overall Study
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812 | 300mg SPN-812 | 400mg SPN-812
Started | 24 | 48 | 50 | 49 | 51
Completed | 21 | 37 | 33 | 35 | 34
Not Completed | 3 | 11 | 17 | 14 | 17
Not completed — Failed to meet eligibility | 0 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 4 | 3 | 1 | 5
Not completed — Lost to Follow-up | 1 | 2 | 5 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 5 | 4 | 4
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Administrative reason | 1 | 0 | 0 | 1 | 0
Not completed — Multiple reasons | 1 | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who were randomized, took at least one dose of study medication, have a baseline Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV) assessment, and have at least one post-baseline ADHD-RS-IV assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812 | 300mg SPN-812 | 400mg SPN-812 | Total
Number analyzed (Participants) | 24 | 45 | 46 | 47 | 44 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (1.89) | 8.2 (1.78) | 9.1 (1.95) | 8.9 (1.95) | 9.0 (2.18) | 8.8 (1.97)
Age, Customized [Count of Participants; unit: Participants]
  6 to 9 years | 16 | 36 | 26 | 30 | 27 | 135
  10 to 12 years | 8 | 9 | 20 | 17 | 17 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 13 | 11 | 13 | 68
  Male | 11 | 27 | 33 | 36 | 31 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 19 | 16 | 22 | 15 | 79
  White | 17 | 22 | 26 | 24 | 28 | 117
  More than one race | 0 | 4 | 1 | 0 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 45 | 46 | 47 | 44 | 206
ADHD RS-IV Total Score [Mean (Standard Deviation); unit: scores on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to the 18 ADHD symptoms per the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV). Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). Total score = sum of 18 items (range: 0 to 54). The higher the score, the more severe the ADHD symptoms (a total score >=26 was an inclusion criterion of this study).
  scores on a scale | 42.4 (7.76) | 42.4 (6.82) | 43.9 (7.45) | 41.3 (7.94) | 40.8 (7.87) | 42.1 (7.57)
ADHD RS-IV Inattention Subscale Score [Mean (Standard Deviation); unit: scores on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to 18 ADHD symptoms per DSM-IV, including 9 items for the Hyperactivity/Impulsivity (HI) subscale and 9 items for the Inattention (IA) subscale. Each item is rated on a 4-point Likert-type scale from (0=never or rarely to 3=very often). The IA Subscale score = sum of all 9 IA items on the ADHD-RS-IV (range:0 to 27). The higher the score, the more severe the IA symptoms of ADHD.
  scores on a scale | 21.9 (4.72) | 22.1 (3.86) | 22.2 (3.57) | 21.8 (3.75) | 21.0 (4.71) | 21.8 (4.06)
ADHD RS-IV Hyperactivity/ Impulsivity Subscale Score [Mean (Standard Deviation); unit: scores on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to 18 ADHD symptoms per DSM-IV, including 9 items for the Hyperactivity/Impulsivity (HI) subscale and 9 items for the Inattention (IA) subscale. Each item is rated on a 4-point Likert-type scale from (0=never or rarely to 3=very often). The HI Subscale score = sum of all 9 HI items on the ADHD-RS-IV (range:0 to 27). The higher the score, the more severe the HI symptoms of ADHD.
  scores on a scale | 20.5 (4.40) | 20.3 (5.15) | 21.7 (5.10) | 19.4 (5.99) | 19.7 (4.43) | 20.3 (5.14)

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of SPN-812 on the Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV)
Description: The Primary Endpoint was the change from baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV) Total score at Week 8 (End of Study). The ADHD-RS-IV is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) symptoms of ADHD. Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). A Total score is calculated by adding the responses of all 18 items (range: 0-54; the higher the score, the more severe the ADHD symptoms). Lower change from baseline scores (<0) represent a better outcome.
Time Frame: Baseline to Week 8 (End of Study)
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who were randomized, took at least one dose of study medication, have a baseline Attention-Deficit/Hyperactivity Disorder Rating Scale, 4th Edition (ADHD-RS-IV) assessment and have at least one post-baseline ADHD-RS-IV assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812 | 300mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 24 | 45 | 46 | 47 | 44
units on a scale | -10.5 (11.82) | -16.7 (14.57) | -18.4 (15.61) | -18.6 (14.38) | -19.0 (14.51)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.0899, ANOVA; Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-13.4 to 1.0]
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.0310, ANOVA; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-15.1 to -0.7]
Statistical Analysis 3: Comparison: Placebo vs 300mg SPN-812; Test type: Superiority; p = 0.0268, ANOVA; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-15.3 to -0.9]
Statistical Analysis 4: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0209, ANOVA; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-15.8 to -1.3]

2. Secondary Outcome: Effect of SPN-812 on Clinical Global Impression - Improvement (CGI-I) Scale
Description: The first additional secondary endpoint was the Clinical Global Impression-Improvement (CGI-I) Scale score at Week 8 (End of Study). The CGI-I scale is a single item assessment of how much the patient's illness has improved or worsened relative to a baseline state prior to the beginning of treatment. The CGI-I is rated on a 7-point Likert scale from 1 to 7, where 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", and 7 = "Very much worse". Successful therapy is indicated by a lower score (<4) in subsequent testing.
Time Frame: Week 8 (End of Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812 | 300mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 24 | 45 | 46 | 47 | 44
units on a scale | 3.0 (0.88) | 2.6 (1.10) | 2.6 (1.26) | 2.2 (1.25) | 2.4 (1.13)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.1305, ANOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.0 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.1376, ANOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.0 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs 300mg SPN-812; Test type: Superiority; p = 0.0090, ANOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.3 to -0.2]
Statistical Analysis 4: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0546, ANOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.1 to 0.0]

3. Secondary Outcome: Effect of SPN-812 on the Clinical Global Impression - Severity (CGI-S) Scale
Description: The second additional secondary endpoint was the change from baseline in the Clinical Global Impression-Severity (CGI-S) Scale score at Week 8 (End of Study). The CGI-S scale is a single item clinician/investigator rating of the clinician's assessment of the severity of the ADHD symptoms in relation to the clinician's total experience with patients with ADHD. The CGI-S was rated on a 7-point Likert scale, where 1 = Normal, not at all ill, 2 = Borderline Ill, 3 = Mildly Ill, 4 = Moderately Ill, 5 = Markedly Ill, 6 = Severely Ill, and 7 = Extremely Ill. Successful therapy is indicated by a lower CGI-S score in subsequent testing. A lower change from baseline score (<0) represents a better outcome.
Time Frame: Baseline to Week 8 (End of Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812 | 300mg SPN-812 | 400mg SPN-812
Number analyzed (Participants) | 24 | 45 | 46 | 47 | 44
units on a scale | -0.8 (0.98) | -1.4 (1.44) | -1.5 (1.44) | -1.6 (1.37) | -1.7 (1.41)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.0708, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.3 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.0309, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.4 to -0.1]
Statistical Analysis 3: Comparison: Placebo vs 300mg SPN-812; Test type: Superiority; p = 0.0148, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.5 to -0.2]
Statistical Analysis 4: Comparison: Placebo vs 400mg SPN-812; Test type: Superiority; p = 0.0136, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.6 to -0.2]

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: Number of subjects is based on the Safety Population (defined as subjects who were randomized and took at least one dose of study medication)
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812 | 300mg SPN-812 | 400mg SPN-812
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/48 | 0/48 | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/48 | 0/48 | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 3/24 | 23/48 | 22/48 | 30/48 | 30/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | 100mg SPN-812 (N=48) | 200mg SPN-812 (N=48) | 300mg SPN-812 (N=48) | 400mg SPN-812 (N=49)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 3 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 5 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 4 | 3 | 5
Fatigue (General disorders) | 0 | 2 | 2 | 1 | 5
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 4
Headache (Nervous system disorders) | 1 | 4 | 6 | 6 | 9
Decreased appetite (Metabolism and nutrition disorders) | 2 | 5 | 7 | 4 | 8
Somnolence (Nervous system disorders) | 1 | 7 | 10 | 11 | 12
Irritability (Psychiatric disorders) | 0 | 1 | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other